CLINICAL TRIAL: NCT01092624
Title: A Randomized, Placebo-Controlled Parallel-Design Trial of the Effect of Solifenacin Treatment for Overactive Bladder in Women With Anterior Vaginal Wall Prolapse Managed With a Pessary (the "PESSARY" Study)
Brief Title: Clinical Trial of Solifenacin Versus Placebo Plus Pessary for Women With Vaginal Prolapse
Acronym: PESSARY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: sponsor closed study due to poor enrollment
Sponsor: Hartford Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TULI003042; VESI-9I04 (Other: Astellas refernce number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-25 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: voiding dysfunction; defecatory dysfunction; vaginal bulge symptoms
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Solifenacin Succinate; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pessary and solifenacin (Experimental)
  Interventions: Drug: Solifenacin; Device: Ring pessary with support, Cooper Surgical, Trumbell, CT Ref # MXPRS03 non-latex
- Pessary and placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Device: Ring pessary with support, Cooper Surgical, Trumbell, CT Ref # MXPRS03 non-latex

INTERVENTIONS:
Drug: Solifenacin — There will be a two-week pessary run-in prior to randomization. If the subject completes the run-in period with no adverse reactions to the pessary, she will come in to the office for a randomization visit. She will be randomized to receive either 5 mg/day (one 5 mg tablet QD) of placebo or 5 mg/day (QD) of solifenacin for 12 weeks. At the end of week 6, patients will be assessed in the office. A standardized medication response questionnaire will be used to assess each subject's response to either the placebo or the solifenacin 5 mg. If the response is not adequate, the dose will be increased. Women whose symptoms have not improved since baseline will have their medication or placebo doses increased to 10 mg daily.
  Other Names: Vesicare
  Arms: Pessary and solifenacin
Drug: Placebo — There will be a two-week pessary run-in prior to randomization. If the subject completes the run-in period with no adverse reactions to the pessary, she will come in to the office for a randomization visit. She will be randomized to receive either 5 mg/day (one 5 mg tablet QD) of placebo or 5 mg/day (QD) of solifenacin for 12 weeks. At the end of week 6, patients will be assessed in the office. A standardized medication response questionnaire will be used to assess each subject's response to either the placebo or the solifenacin 5 mg. If the response is not adequate, the dose will be increased. Women whose symptoms have not improved since baseline will have their medication or placebo doses increased to 10 mg daily.
  Arms: Pessary and placebo
Device: Ring pessary with support, Cooper Surgical, Trumbell, CT Ref # MXPRS03 non-latex — There will be a two-week pessary run-in prior to randomization. If the subject completes the run-in period with no adverse reactions to the pessary, she will come in to the office for a randomization visit. She will be randomized to receive either 5 mg/day (one 5 mg tablet QD) of placebo or 5 mg/day (QD) of solifenacin for 12 weeks. At the end of week 6, patients will be assessed in the office. A standardized medication response questionnaire will be used to assess each subject's response to either the placebo or the solifenacin 5 mg. If the response is not adequate, the dose will be increased. Women whose symptoms have not improved since baseline will have their medication or placebo doses increased to 10 mg daily.

SUMMARY:
This study will evaluate the effect of pessary therapy, with and without Solifenacin (Vesicare), on symptoms of over active bladder and bladder function in women with overactive bladder symptoms and pelvic organ prolapse.

Study Hypotheses:

Null hypothesis, HO: Reduction of anterior vaginal wall prolapse and treatment with solifenacin does not improve overactive bladder symptoms more than reduction of anterior vaginal wall prolapse and placebo.

Alternate hypothesis, HA: Reduction of anterior vaginal wall prolapse and treatment with solifenacin does improve overactive bladder symptoms more than reduction of anterior vaginal wall prolapse and placebo.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) affects approximately half of all women over age 501. The most common type of POP is anterior vaginal wall prolapse. Symptoms associated with POP include: voiding dysfunction, defecatory dysfunction and vaginal bulge symptoms. Treatments for pelvic organ prolapse include among other options, vaginal pessary or surgery. Several studies have documented improved vaginal bulge symptoms in women treated with a pessary2,3,4; however, data are sparse regarding the effect of pessaries on lower urinary tract symptoms, specifically with regard to over active bladder symptoms.

Overactive bladder, observed in approximately 40% of women 50 years of age or older, is very common in women with pelvic organ prolapse. Two retrospective studies have shown improvement in women with overactive bladder symptoms following treatment with a vaginal pessary. One study (using a non-validated questionnaire) found that, at two month follow-up, patients successfully fitted with a pessary experienced a reduction in slightly less than half of their urge incontinence symptoms.5 A second study (using the Sheffield pelvic organ prolapse symptom questionnaire), revealed that 4 months after insertion of a pessary, 38% of patients experienced reduced urinary urgency, and 29% experienced reduced urge urinary incontinence6. Despite these data, many women stop using a pessary secondary to complaints of increased urine incontinence. More information is needed on pessary therapy impact on bladder function.

Specific Aim(s):

This study will prospectively evaluate women with pelvic organ prolapse and overactive bladder symptoms treated with either

1. a pessary and solifenacin, or
2. a pessary and placebo. We will assess the effects of these therapies on overactive bladder symptoms over the course of the 14-week study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* Have experienced symptoms of overactive bladder (e.g., urinary urgency, frequency, or urge incontinence) for at least 3 months. Specifically women must average 8 or more voids in 24 hours and have 3 or more episodes of urinary urgency or urge incontinence over the 72 hours when the diary is being completed.
* A practitioner trained in the pelvic organ prolapse quantification examination will evaluate each woman's pelvic organ support and vaginal dimensions. Women with a stage 1 or greater vaginal prolapse will be eligible for the study.

Exclusion Criteria:

* The presence of factors that would contraindicate use of antimuscarinic medications (e.g. urine retention, narrow angle glaucoma, uncontrolled constipation, dementia)
* An existing condition that would contraindicate use of a vaginal pessary (e.g., patient's vaginal length <6 cm)
* Patient is currently using a vaginal pessary.
* Patient is unable to tolerate an object in vagina
* Patient has a history of cervical, vaginal or endometrial cancer
* Patient is not able to speak English
* Patient is currently using an anticholinergic medication, or has used one in the past 30 days
* Patients with mixed urine incontinence that is predominantly stress urine incontinence (determined by their baseline PFDI)
* Patients with a known allergy to solifenacin.
* Patients with severe hepatic impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The Effect of These Therapies on Over-Active Bladder Symptoms | 14-Weeks
  Using the PFDI and PFIQ and a standardized medication response questionnaire to assess each subject's response to either the placebo or the solinefacin at Week 6 and Week 14, we will evaluate the effect of these therapies on subjects' bladder symptoms over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tulikangas, MD, Principal Investigator — Hartford Hospital, Women's Specialty Services
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States